CLINICAL TRIAL: NCT02808247
Title: A Phase II Multicenter Study Comparing the Efficacy of the Oral Angiogenesis Inhibitor Nintedanib With the Intravenous Cytotoxic Compound Ifosfamide for Treatment of Patients With Advanced Metastatic Soft Tissue Sarcoma After Failure of Systemic Non-oxazaphosporine-based First Line Chemotherapy for Inoperable Disease "ANITA"
Brief Title: Ph II Nintedanib vs. Ifosfamide in Soft Tissue Sarcoma
Acronym: ANITA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Exceed of pre-specified number of failures in the experimental arm
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1506-STBSG; 2016-002093-12 (EudraCT Number)
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Sarcoma, Soft Tissue
Keywords: advanced metastatic soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — nintedanib; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (arm A): Nintedanib (Experimental): Nintedanib 200 mg twice daily orally. Nintedanib will be given continuously until clinically relevant disease progression according to the investigator's assessment or until other criteria for treatment discontinuation are met as specified in the protocol. Dosing beyond RECIST 1.1 progression is allowed for the oral agent if the patient still derives benefit from the treatment.
  Interventions: Drug: Nintedanib
- Standard arm (arm B): Ifosfamide (Active Comparator): Ifosfamide 3 g/m2 intravenously on days 1, 2 and 3 every 21 days for up to a maximum of 6 cycles.
  Interventions: Drug: Ifosfamide

INTERVENTIONS:
Drug: Nintedanib — Pharmaceutical form: Soft gelatine capsule Pharmaceutical code: Nintedanib (BIBF1120) Source: Boehringer Ingelheim Pharma GmbH & Co. KG Unit strength: 100 mg and 150 mg capsules Daily dose: 400 mg (200 mg twice daily p.o.) Route of administration: oral
  Other Names: BIBF1120
  Arms: Experimental arm (arm A): Nintedanib
Drug: Ifosfamide — Ifosfamide will be given at a dose of 3 g/m2 intravenously on days 1, 2 and 3 every 21 days. The total dose per cycle is 9 g/m2
  Arms: Standard arm (arm B): Ifosfamide

SUMMARY:
This is a prospective, multicentric, randomized, open label Phase II trial investigating whether the oral angiogenesis inhibitor nintedanib, as compared to the intravenous cytotoxic compound ifosfamide, given for patients with advanced, inoperable and/or metastatic STS after failure of first line chemotherapy prolongs progression-free survival.

The primary objective of the trial is to evaluate whether nintedanib given as second-line therapy for advanced, inoperable and/or metastatic STS prolongs progression-free survival when compared with ifosfamide.

Secondary objectives are to evaluate the efficacy of nintedanib as compared to ifosfamide in terms of progression-free survival rate at 12 weeks, overall survival, objective response rate, patient benefit rate, response duration, total duration of treatment with nintedanib safety, Health related Quality of Life and Health Economics.

Exploratory objectives include an analysis of putative predictive biomarkers for the anti-tumor effects of the investigational agent nintedanib.treatment.

ELIGIBILITY:
Inclusion Criteria/Exclusion Criteria:

* Histologically proven advanced, inoperable and/or metastatic malignant STS of intermediate or high grade, excluding the:
* Well-differentiated liposarcoma/atypical lipoma
* Embryonal rhabdomyosarcoma
* Chondrosarcoma (extraskeletal myxoid chondrosarcoma is eligible)
* Osteosarcoma (extraskeletal osteosarcoma is eligible)
* Ewing family of tumors/primitive neuroectodermal tumor
* Gastro-intestinal stromal tumor
* Dermatofibrosarcoma protuberans
* For STS where no established grading system exists, or sarcoma subtypes which are very indolent or have an unpredictable clinical behavior, patient entry requires prospective approval in writing, on a case-by-case basis by the Study Coordinator of this trial and EORTC Headquarters (HQ).
* Representative formalin fixed, paraffin embedded tumor blocks or unstained tissue slides, either from the primary tumor or a metastatic lesion, must be available for histological central review. Histological central review is not required before treatment start but it is mandatory to send unstained tumor slides (blocks optional) at time of study entry. Local histopathological diagnosis will be accepted for entry into this trial.
* Prior to study enrolment, all patients need to have confirmed RECIST 1.1 disease progression based on local investigator's assessment.
* Presence of measurable disease according to RECIST 1.1.
* Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are considered non-measurable unless there has been demonstrated progression (20 % increase) in the assessed lesion since the local treatment.
* No radiographic evidence of cavitary lesions (either primary tumor or metastatic lesions).
* No centrally located tumors with radiographic evidence of local invasion of major blood vessels.
* No history of central nervous system metastasis or leptomeningeal tumor spread.
* No active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month before randomization).
* One (and no less or more than one) line of previous systemic chemotherapy for advanced, inoperable and/or metastatic malignant STS.
* Prior neoadjuvant, adjuvant and or first-line maintenance systemic chemotherapy for locally advanced or metastatic STS is allowed and does count as zero lines of treatment, provided that the disease did not progress during neoadjuvant and/or adjuvant therapy or within 12 weeks after completion of the perioperative treatment. In case the disease progressed during neoadjuvant, adjuvant and or first-line maintenance systemic chemotherapy or within 12 weeks after its completion, the treatment is counted as one line and the patient can theoretically participate in the trial, provided all other selection criteria are met.
* No prior exposure to an oxazaphosphorine agent, including but not limited to ifosfamide, cyclophosphamide, trofosfamide or evofosfamide (TH-302).
* No prior exposure to oral or intravenous angiogenesis inhibitors, including but not limited to tyrosine kinase inhibitors such as pazopanib, sunitinib, sorafenib, axitinib or similar or monoclonal antibodies targeting angiogenesis.
* No other anti-cancer therapy (systemic therapy, radiotherapy (except for brain and extremities), surgery, limb perfusion, immunotherapy) within 28 days prior to randomization.
* No treatment with another investigational agent within 28 days prior to randomization.
* No treatment with another investigational agent concomitantly with the trial.
* No known hypersensitivity to or known specific contraindications for the use of nintedanib or ifosfamide.
* No known hypersensitivity to peanut or soy bean.
* Age 18 years or older.
* WHO performance status (PS) 0-2.
* Life expectancy of at least 3 months.
* Adequate bone marrow, liver and renal function and coagulation parameters:
* neutrophils ≥ 1.5 x 109/L;
* hemoglobin ≥ 9 g/dL (or ≥ 5.6 mmol/L). Blood transfusions or the administration of hematopoietic growth factors are allowed to achieve these baseline values;
* platelets ≥ 100 x 109/L. Platelet transfusions or the administration of hematopoietic growth factors are allowed to achieve these baseline values;
* Total bilirubin ≤ ULN;
* Patients with Gilbert syndrome and/or bilirubin < 2xULN and normal AST/ALT are eligible;
* SGPT/ALT and SGOT/AST ≤ 2.5 x ULN for patients with liver metastasis;
* SGPT/ALT and SGOT/ AST ≤ 1.5x ULN for patients without liver metastasis;
* Serum creatinine or creatinine clearance/eGFR within normal limits to baseline, assessed as per local standard method;
* No proteinuria CTCAE grade 2 or greater;
* International normalized ratio (INR) ≤ 2;
* Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 50% of institutional ULN.
* No Child Pugh B or C hepatic impairment.
* Normal cardiac function (left ventricular ejection fraction (LVEF) assessed by multi-gated acquisition scan or cardiac ultrasound within normal range of the institution), 12 lead electrocardiogram (ECG) without clinically relevant abnormalities. No Class III or IV congestive heart failure, angina pectoris, myocardial infarction within 1 year before registration/randomization, clinically significant cardiac arrhythmia or pericardial effusion.
* No uncontrolled arterial hypertension defined at baseline as blood pressure ≥ 150/100 mmHg despite adequate medical therapy.
* No use of therapeutic anticoagulation (except low-dose heparin and/or heparin flush as needed for maintenance of an indwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325 mg per day).
* No known inherited predisposition for bleeding or thromboembolism.
* No history of clinically significant hemorrhagic or thromboembolic event in the past 6 months.
* Absence of active or uncontrolled infections in particular if requiring systemic antibiotics or antimicrobial therapy.
* No previous encephalopathy of any cause or other significant neurological condition.
* No acute or chronic, clinically relevant inflammation of urinary bladder.
* Absence of serious illnesses or medical conditions, including a history of chronic alcohol abuse, active and chronic hepatitis B or C, chronic infection with HIV or clinically relevant liver cirrhosis.
* Absence of active gastrointestinal disorders or abnormalities that interfere with absorption of the study drug.
* No major injuries and/or surgery within the past 28 days prior to randomization with incomplete wound healing and/or planned surgery during the on-treatment study period.
* No persistence of clinically relevant therapy-related toxicity from previous chemotherapy and/or radiotherapy. Grade 1 or 2 adverse events (AEs) are acceptable.
* No history, within the past five years, of malignancies other than STS (except: basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix, resected prostate cancer staged pT1-2 with Gleason Score ≤ 6 and postoperative PSA < 0.5 ng/ml). Patients with a history of other malignancies who are disease-free from that condition for more than 5 years are eligible.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration/randomization in the trial.
* No active alcohol or drug abuse.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to randomization.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 3 months (nindetanib) and 6 months (ifosfamide) after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly. Since the effect of nintedanib on the metabolism and efficacy of contraceptives has not been investigated, barrier methods should be applied as a second form of contraception, to avoid pregnancy.
* Female subjects who are breast feeding should discontinue nursing prior to randomization and until 6 months after the last study treatment.
* Sexually active male participants must use a barrier method of contraception (e.g., condom) during the study treatment period and for at least 3 months after the last study treatment.
* Before patient registration/randomization, written informed consent must be obtained according to international conference on harmonisation/Good clinical practice (ICH/GCP) and national/local regulations.
* Patients can only be randomized in this trial once. Important note: All eligibility criteria must be adhered to, in case of potential deviation a discussion with EORTC Headquarters and study coordinator is mandatory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 4 years from first patient in
  progression-free survival (PFS) defined according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival rate at 12 weeks (binary) | 4 years from first patient in
Overall survival | 4 years from first patient in
Objective response rate | 4 years from first patient in
  Objective tumor response as defined by RECIST 1.1
Clinical benefit rate | 4 years from first patient in
Response duration | 4 years from first patient in
  Duration of response will be measured for patients achieving an objective response
Total duration of treatment with nintedanib (including treatment beyond RECIST progression) | 4 years from first patient in
Safety (Common Toxicity Criteria CTCAE 4.0) | 4 years from first patient in
Health related quality of life (QLQ-C30) | 4 years from first patient in
  Quality of life will be assessed with the EORTC QoL Questionnaire (QLQ-C30) version 3.0
Health economics (EQ-5D-5L, health care resource utilities) | 4 years from first patient in
  Patient reported utility: EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoeffski, MD, Principal Investigator — U.Z. Leuven - Campus Gasthuisberg (147)
Locations (13):
- Belgium (3):
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc (121), Brussels
  - U.Z. Leuven - Campus Gasthuisberg (147), Leuven
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard (227), Lyon
  - Gustave Roussy (225), Villejuif
- Vilnius University Hospital Santariskiu Santaros Clinics Klinikos (9453), Vilnius, Lithuania
- Netherlands (2):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis (301), Amsterdam
  - Leiden University Medical Centre (310), Leiden
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- Spain (2):
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Barcelona
  - Hospital Universitario San Carlos (366), Madrid
- Royal Marsden Hospital - Chelsea, London (613), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schoffski P, Toulmonde M, Estival A, Marquina G, Dudzisz-Sledz M, Brahmi M, Steeghs N, Karavasilis V, de Haan J, Wozniak A, Cousin S, Domenech M, Bovee JVMG, Charon-Barra C, Marreaud S, Litiere S, De Meulemeester L, Olungu C, Gelderblom H. Randomised phase 2 study comparing the efficacy and safety of the oral tyrosine kinase inhibitor nintedanib with single agent ifosfamide in patients with advanced, inoperable, metastatic soft tissue sarcoma after failure of first-line chemotherapy: EORTC-1506-STBSG "ANITA". Eur J Cancer. 2021 Jul;152:26-40. doi: 10.1016/j.ejca.2021.04.015. Epub 2021 May 29. PMID 34062484